CLINICAL TRIAL: NCT02075684
Title: Office-based Percutaneous Ultrasound-guided Renal Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of Michigan (Other); University of California, Los Angeles (Other); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Jaime Landman, Professor of Urology and Radiology, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20139312
Record Dates: First submitted 2013-08-21; First posted 2014-03-03 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Renal Cortical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- In-office, Percutaneous Renal Biopsy (Other)
  Interventions: Procedure: Renal Biopsy

INTERVENTIONS:
Procedure: Renal Biopsy

SUMMARY:
The purpose of this research study is to create a prospectively maintained, multicenter database of patients undergoing renal biopsy for renal masses performed percutaneously (through skin), via an 18 gauge biopsy needle (.048 inches). In this database, the investigators will collect and maintain the data from the biopsy procedure. This will allow us to evaluate our experience with this procedure as well as to participate in multi-institutional collaborative studies in the future. At University of California Irvine, the investigators routinely biopsy patients with renal masses under real-time ultrasound control. Percutaneous renal biopsy under ultrasound guidance is a routine procedure performed to diagnose renal mass histopathology. The safety and efficacy of this procedure has been well documented in the literature. The indications for percutaneous renal biopsy have expanded as there has been a substantial increase in the number of renal masses that are being diagnosed, and the acceptance of percutaneous biopsy continues to expand in parallel. The biopsy procedure is part of your normal standard of care and if not being done for this research project.

ELIGIBILITY:
Inclusion Criteria:

* Must be undergoing standard percutaneous renal biopsy
* Patients must be ≥18 years of age
* Must be able to understand and render voluntary, written informed consent

Exclusion Criteria:

* Patients <18 years of age
* Pregnant women
* Coagulopathy
* Active urinary tract infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2024-04 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Tumor Characteristics | Baseline
  Tumor characteristics will be recorded at Baseline (from preoperative imaging) using the R.E.N.A.L. Nephrometry scoring system which captures tumor radius (R), depth within renal parenchyma (E), nearness to collecting system (N), anterior/posterior location (A) and polarity (L).

SECONDARY OUTCOMES:
Verbal analog pain scale | Baseline, 1 hour post procedure, and 3 days - 3 weeks post-procedure
  Preprocedural and postprocedure verbal analog pain scale. Verbal analog pain scale (0 to 10) will be recorded immediately after and 60 minutes after the procedure. Additional pain assessment will be performed at a follow-up visit 3 days to 3 weeks after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Landman, MD, Principal Investigator — UCI Health Department of Urology
Locations (1):
- Universty of California Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not intend to release individual data to other researchers.

REFERENCES:
- See also: Related Info — http://research.uci.edu